CLINICAL TRIAL: NCT02968576
Title: Bioequivalence of Tenofovir and Emtricitabine Following Overencapsulation
Acronym: A-TEAM
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Colorado, Denver (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Basic Science
Other Study IDs: 16-1478
Record Dates: First submitted 2016-11-08; First posted 2016-11-18 (Estimated); Results first posted 2019-05-14 (Actual); Last update posted 2020-03-06 (Actual); Status verified 2020-02

CONDITIONS: Healthy Volunteers; Pharmacokinetics
Keywords: healthy volunteers; pharmacokinetics
MeSH Terms: interventions — Tenofovir; Emtricitabine; Tablets; Emtricitabine, Tenofovir Disoproxil Fumarate Drug Combination

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Truvada (Active Comparator): Naked form Truvada (drug)
  Interventions: Drug: TENOFOVIR DISOPROXIL FUMARATE 300 Mg / EMTRICITABINE 200 Mg ORAL TABLET [TRUVADA]
- PSS-Truvada (Experimental): Proteus Sensor System (PSS) (device) encapsulated Truvada (drug)
  Interventions: Drug: TENOFOVIR DISOPROXIL FUMARATE 300 Mg / EMTRICITABINE 200 Mg ORAL TABLET [TRUVADA]; Device: Proteus Sensor System

INTERVENTIONS:
Drug: TENOFOVIR DISOPROXIL FUMARATE 300 Mg / EMTRICITABINE 200 Mg ORAL TABLET [TRUVADA]
  Other Names: Truvada
Device: Proteus Sensor System
  Other Names: PSS
  Arms: PSS-Truvada

SUMMARY:
Poor adherence to tenofovir (TDF) and emtricitabine (FTC) for Human Immunodeficiency Virus (HIV) pre-exposure prophylaxis (PrEP) is common and the leading cause of therapeutic failure. The investigators need better ways to measure adherence in patients on PrEP. This application will address the need to measure adherence by evaluating an integrated technology system, Proteus Discover, when combined with Truvada. The Proteus Sensor System (PSS) will confirm that Truvada was taken, monitor adherence in both recent and long term dosing, and provides feedback to encourage adherence. The goal of this study is to determine whether the use of the PSS with Truvada will vary the drug concentrations of FTC/TDF. Participants will have 2 study visits where they will be randomized to either start with the combined PSS with Truvada or just Truvada alone. Study participants will come to the Clinical & Translational Research Center (CTRC) in the morning and take the assigned dose and will then have blood drawn at about .25, 0.5, 1, 2, 4, 6, and 10 hours after medication is taken. Participants will then return to the CTRC for blood draws 24, 48, and 72 hours after they took the dose on the first day. The second visit will mimic the first except that the participant will take the other dose form.

ELIGIBILITY:
Inclusion Criteria:

1. Ambulatory 18-45 year old adults.
2. Ability to comply with study procedures

Exclusion Criteria:

1. Inability to give informed consent
2. Pregnancy or planning to become pregnant within 3 months of study completion
3. Currently breastfeeding
4. High risk of HIV-1 infection (for example: sexually active with an HIV infected partner; men who have sex with men who may engage in condom-less intercourse with HIV-infected partners or partner of unknown status during the study; males or females who exchange sex for money, shelter, or gifts; active injection drug use or during the last 12 months; newly diagnosed sexually transmitted infections in last 6 months)
5. Positive HIV+ ELISA or suspected acute HIV infection in the opinion of the clinician. (example signs and symptoms of acute HIV infection include combinations of fever, headache, fatigue, arthralgia, vomiting, myalgia, diarrhea, pharyngitis, rash, night sweats, and adenopathy cervical or inguinal)
6. Positive hepatitis B virus (HBV) surface antigen test.
7. Uncontrolled or symptomatic bone disease or history of non-traumatic bone fractures
8. Active psychiatric illness or alcohol/drug abuse that, in the opinion of the investigators, would interfere with study requirements
9. Creatinine clearance < 60 ml/min, or history of serious renal disease
10. Urine dipstick protein ≥ 2+
11. Total bilirubin and/or hepatic transaminases (ALT and AST) ≥ 2.5x upper limit of normal
12. Absolute neutrophil count ≤ 1,500/mm3, platelets count ≤ 100,000/mm3, or hemoglobin ≤ 10 g/dL.
13. Any laboratory value or uncontrolled medical conditions that, in the opinion of investigators, would interfere with the study conditions or increase risk to the participant
14. > Grade I abnormalities in screening laboratory tests (Complete Blood Count, Comprehensive Metabolic Panel, Lipase, Phosphorus) per Division of AIDS (DAIDS) Grading Table
15. Contraindicated concomitant medications based upon product information or that, in the opinion of the investigators, would interact with the study medications or increase risk to participant such as: investigational agents (within 30 days of enrollment), aminoglycosides, ganciclovir/valganciclovir, chronic high-dose acyclovir/valacyclovir (>800mg acyclovir or > 500mg valacyclovir for > 7 days), cyclosporine, amphotericin B, foscarnet, and cidofovir, and products with same or similar active ingredients as the study medications including TRUVADA®, ATRIPLA®, COMPLERA®, EMTRIVA®, VIREAD®; or drugs containing lamivudine or adefovir, which are close analogs of FTC and tenofovir.
16. Current participation in other interventional research studies

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 25 (Actual)
Dates: Start 2016-12 (Actual); Primary Completion 2017-04 (Actual); Study Completion 2017-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Peter Anderson, PharmD, Principal Investigator — University of Colorado, Denver

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Ibrahim ME, Brooks KM, Castillo-Mancilla JR, McHugh C, Morrow M, Brothers J, MaWhinney S, Hosek S, Huhn G, Anderson PL. Short Communication: Bioequivalence of Tenofovir and Emtricitabine After Coencapsulation with the Proteus Ingestible Sensor. AIDS Res Hum Retroviruses. 2018 Oct;34(10):835-837. doi: 10.1089/AID.2018.0081. Epub 2018 Sep 5. PMID 30047286

RESULTS

PARTICIPANT FLOW:
Recruitment Details: IRB approval was obtained for 48 subjects to allow for screen failures, withdrawals, lost to follow up, etc.
Groups:
- Truvada First, Then Coencapsulated PSS-Truvada: Single dose of unencapsulated Truvada (Tenofovir disoproxil fumarate 300mg/Emtricitabine 200mg), 14-day washout followed by single dose of Truvada coencapsulated with the Proteus Sensor System (PSS) (device).
- Coencapsulated PSS-Truvada First, Then Truvada: Single dose of Truvada (Tenofovir disoproxil fumarate 300mg/Emtricitabine 200mg) coencapsulated with the Proteus Sensor System (PSS) (device), 14-day washout followed by single dose of unencapsulated Truvada.
Period: Overall Study
Arm/Group | Truvada First, Then Coencapsulated PSS-Truvada | Coencapsulated PSS-Truvada First, Then Truvada
Started | 11 | 14
Completed | 11 | 13
Not Completed | 0 | 1
Not completed — Pregnancy | 0 | 1

BASELINE CHARACTERISTICS:
Groups:
- All Participants: Single dose of unencapsulated and coencapsulated TDF/FTC. A 14-day washout separated each dosing.
Arm/Group | All Participants
Number analyzed (Participants) | 25
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 25
  >=65 years | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 14
  Male | 11
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Race/Ethnicity: Hispanic | 3
  Race/Ethnicity: African American | 3
  Race/Ethnicity: Caucasian | 19

OUTCOME MEASURES:

1. Primary Outcome: Peak Plasma Concentration (Cmax)
Description: Tenofovir and emtricitabine concentration max (Cmax) following FTC/TDF in the overencapsulated versus non-encapsulated form. Drug concentrations will be assayed with validated liquid chromatography tandem mass spectrometry (LC-MS/MS) methodology.
Time Frame: 0, 1, 2, 3, 4, 6, 8, 12, 24, 48, 72, 96 hours post-dose
Population: All subjects who completed the study: single dose of unencapsulated and coencapsulated TDF/FTC. A 14-day washout separated each dosing.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng/mL
Units Other Than Participants: PK timepoint samples
Arm/Group | All Participants
Number analyzed (Participants) | 24
Number analyzed (PK timepoint samples) | 477
ng/mL
  TFV Cmax-unencapsulated | 222 (37)
  TFV Cmax-coencapsulated | 229 (32)
  FTC Cmax-unencapsulated | 1567 (33)
  FTC Cmax-coencapsulated | 1684 (29)

2. Primary Outcome: Area Under the Concentration-time Curve (AUC)
Description: Tenofovir and emtricitabine area under the concentration-time curve (AUC) following FTC/TDF in the overencapsulated versus non-encapsulated form. Drug concentrations will be assayed with validated liquid chromatography tandem mass spectrometry (LC-MS/MS) methodology.
Time Frame: 0, 1, 2, 3, 4, 6, 8, 12, 24, 48, 72, 96 hours post-dose
Population: as for outcome 1
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng*h/mL
Units Other Than Participants: PK timepoint samples
Arm/Group | All Participants
Number analyzed (Participants) | 24
Number analyzed (PK timepoint samples) | 477
ng*h/mL
  TFV AUC-unencapsulated | 1978 (27)
  TFV AUC-coencapsulated | 2042 (26)
  FTC AUC-unencapsulated | 9342 (23)
  FTC AUC-coencapsulated | 9512 (20)

ADVERSE EVENTS:
Time Frame: Time of consenting to study exit, Max. 54 days
Description: AEs were graded per the DAIDS Table for Grading the Severity of Adult and Pediatric Adverse Events, Version 2.0, November, 2014. Available on the DAIDS RSC Web site: http://rsc.tech-res.com/safetyandpharmacovigilance/
Groups:
- All Subjects: Overall, the study showed an unremarkable and expected AE profile. At study initiation Truvada was FDA approved thus, the AE profile was already established. This study was not designed to collect new safety data or to update the established AE/Safety profiles for Truvada. Therefore AE data was combined for all dosing regimens since AEs reported per arm/group are not meaningful for research or clinical applications.
Arm/Group | All Subjects
All-Cause Mortality (participants affected / at risk) | 0/25
Serious Adverse Events (participants affected / at risk) | 0/25
Other Adverse Events (participants affected / at risk) | 14/25
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | All Subjects (N=25)
Nausea (Gastrointestinal disorders) | 3 (3)
Vomitting (Gastrointestinal disorders) | 1 (1)
Headache (General disorders) | 1 (1)
Common Cold (General disorders) | 7 (7)
Respiratory Infection (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Facial Swelling (General disorders) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2016-09-21): https://cdn.clinicaltrials.gov/large-docs/76/NCT02968576/Prot_SAP_000.pdf